CLINICAL TRIAL: NCT07105397
Title: Evaluating Conversational Artificial Intelligence for Depression Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00000316; ME-2024C1-36732 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2025-07-01; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: major depression; antidepressant; large language model; conversational agent; artificial intelligence; AI; NLP; major depressive disorder; medical record augmented generation; patient simulation; testbed
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: In this randomized controlled trial, patients will be randomly exposed to two comparators: the conversational intake and a structured questionnaire intake.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Structured Survey Questionnaire (Active Comparator): Participants complete a structured, multiple-choice questionnaire designed to efficiently collect medical history. This intake method uses decision trees to sequentially select questions based on prior responses, maximizing information gain and minimizing unnecessary queries. The questionnaire systematically gathers patient demographics, depression history, and previous antidepressant use through closed-ended, mutually exclusive, and exhaustive response options.
  Interventions: Other: Structured Survey Questionnaire
- Conversational AI system (Experimental): Participants engage in medical history intake through an interactive conversational AI system designed to create patient-centered interactions. The system utilizes advanced Large Language Models (LLMs) to understand patient inputs, interpret context, and generate coherent, natural language responses with an empathetic tone. Within the conversational AI, a Dialogue Manager guides the conversation by prioritizing medically relevant topics, ensuring efficient data collection and minimizing off-topic dialogue. To enhance patient safety, conversations are continuously monitored in real-time by trained human-in-the-loop monitors, who can promptly intervene if potential safety risks, such as indications of self-harm, are identified. The primary intent of the conversational AI system is to streamline the antidepressant recommendation process, provide personalized patient interactions, and foster patient comfort and therapeutic alliance through empathetically toned responses.
  Interventions: Other: Conversational AI system

INTERVENTIONS:
Other: Conversational AI system — The conversational AI intervention utilizes interactive dialogue to collect patient medical histories. Powered by advanced Large Language Models (LLMs), the system engages participants in open-ended, natural language conversations. A Dialogue Manager coordinates the dialogue, ensuring conversations remain medically relevant, personalized, and safe. Clinicians monitor the interactions in real-time, validating and ensuring accuracy of antidepressant recommendations informed by an evidence-based Antidepressant Knowledgebase.
  Arms: Conversational AI system
Other: Structured Survey Questionnaire — The structured questionnaire intake utilizes a predefined, multiple-choice survey that systematically collects patient medical history without conversational interaction. Questions are algorithmically selected based on the patient's earlier responses to maximize information efficiency, typically requiring fewer than 13 items. Patients select from standardized responses (including options like "I do not know" or "I do not want to say"). Contextual help messages are provided as needed. Upon completion, the system generates antidepressant recommendations using the same Antidepressant Knowledgebase as the Conversational AI system, clearly explaining its rationale. A prototype version is available at http://MeAgainMeds.com, with ongoing development to enhance features and usability.
  Arms: Structured Survey Questionnaire

SUMMARY:
The goal of this clinical trial is to evaluate how a conversational method of collecting medical history affects patients' perceptions and experiences compared to traditional online, closed-ended surveys. Both methods collect identical medical history information, can be completed by patients at home, and do not disrupt routine clinical care.

The primary questions this study aims to answer are:

1. Does conversational intake affect patients' perceptions of empathy during their clinical interactions?
2. Does conversational intake strengthen the therapeutic bond patients feel toward their clinicians compared to traditional surveys?

Participants will be randomly assigned to one of two intake methods:

1. Conversational intake: Participants answer questions about their medical history through a natural, dialogue-based interface.
2. Closed-ended survey intake: Participants complete a structured, multiple-choice questionnaire about their medical history.

After completing their assigned intake method, participants will rate their experience, particularly in terms of empathy and therapeutic bond, and compare it to their usual interactions with their own clinicians.

DETAILED DESCRIPTION:
Conversational artificial intelligence (AI) systems, such as those based on Large Language Models (LLMs) like ChatGPT, offer innovative ways to engage patients in health-related conversations. Despite these advances, challenges remain regarding patient safety and system reliability. Specific concerns include biased recommendations against certain patient groups, inaccuracies or misleading responses, and mechanical, unempathic interactions, particularly during sensitive moments such as when patients express suicidal thoughts. Testing conversational AI in healthcare settings is complicated due to the diverse medical, linguistic, and behavioral characteristics exhibited by patients.

This study addresses these challenges by developing an advanced conversational AI system guided by a structured knowledge-based topic network to maintain conversation relevance and coherence. Additionally, the investigators introduce a novel patient simulator methodology that mimics diverse medical histories, linguistic styles, and behavioral interactions, enhancing pre-clinical testing rigor.

The research focuses specifically on the clinical context of depression management, aiming to optimize antidepressant selection. Currently, many patients undergo a frustrating and costly trial-and-error process to find effective antidepressants. The study compares two approaches designed to streamline and personalize this process:

1. Conversational AI Intake: Engages patients through flexible, open-ended dialogue to gather medical history and generate personalized antidepressant recommendations.
2. Structured Questionnaire Intake: Utilizes a closed-ended, multiple-choice format to systematically collect patient medical histories for antidepressant recommendation.

Both methods leverage a curated, evidence-based knowledgebase of 15 commonly used antidepressants, considering factors like patient age, gender, comorbidities, and previous antidepressant use. The accuracy and completeness of the AI-generated recommendations are rigorously verified in by clinicians prior to any medication changes, adhering to FDA safety requirements.

A primary goal of the project is to evaluate how conversational AI impacts patient-centered outcomes, specifically patient perceptions of empathy, therapeutic bond, and communication quality. Patients with major depressive disorder will be recruited online, enhancing participant diversity and representativeness. Participants will be randomly assigned to either the conversational AI or the structured questionnaire method. Outcomes will include differences in data completeness, patient perceptions of empathy, and strength of therapeutic alliance.

Beyond immediate clinical outcomes, the project's methodological advancements, particularly the development of robust, bias-mitigated conversational systems and comprehensive patient simulation for AI testing, will have broad applicability across healthcare domains. The conversational AI and patient simulator will be made publicly available at no cost, providing tools that other researchers, clinicians, and healthcare providers can utilize and adapt to various health contexts.

Patient and stakeholder engagement is integral to the study. A representative advisory board, including patients with lived experience of depression, clinicians, mental health advocates, and researchers, guides all phases of the project. This collaborative framework ensures that the research remains patient-centered and responsive to real-world clinical needs and experiences.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 85 years old
* have a major depression diagnosis from a clinician and score 10 or higher on the Patient Health Questionnaire (PHQ-9)
* reside in a state where study clinicians are licensed
* have access to the Internet via phone or computer
* have no language, sensorial, or cognitive barriers to providing written informed consent
* must have a primary care provider, a mental health specialist, or agree to see a study clinician

Exclusion Criteria:

- has clinically diagnosed bipolar disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2028-04-15 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Perceptions of empathy | From enrollment up to 4 months after participation
  The primary outcome assesses the impact of intake methods (conversational AI vs. structured survey) on patients' perceptions of empathy. Patient empathy perceptions will be measured using the Jefferson Scale of Empathy (JSE), a validated instrument. A higher JSE score means higher perceptions of empathy. We hypothesize that patients interacting with the conversational AI will report higher perceived empathy scores compared to those using the structured survey. Data analysis will employ comparison of independent means through Analysis of Variance (ANOVA). If randomization does not yield comparable groups, we will apply covariate-balanced ANOVA. Power analysis (conducted in RStudio) indicated a sample size of 130 patients (power = 0.80, significance level = 0.05), based on a mean JSE score of 116.6, standard deviation of 10.56, and an assumed medium effect size (5% mean difference).

SECONDARY OUTCOMES:
Communication Accommodation | From enrollment up to 4 months after participation
  We will assess communication accommodation to determine whether the conversational AI meets patient needs through a content analysis of conversation transcripts. This analysis will rate three key dimensions: empathy, communication quality, and effectiveness. Codes for each are drawn from validated, widely used scales. From this, we will generate composite scores to classify AI conversations as high or low in each dimension and overall. To validate our findings, we will compare content analysis scores with patient self-reports on perceived levels (high or low) of empathy, quality, and effectiveness. Together, these data will provide a robust evaluation of the AI's communication accommodation.
Therapeutic Alliance Between System and Patient | From enrollment up to 4 months after participation
  We will use a multi-measure strategy to evaluate the therapeutic alliance between the AI system and patients. This includes four related measures. First, a content analysis of patient-AI conversation transcripts will rate the level of empathy using a validated scale from prior studies. These ratings will generate a score classifying each conversation as high or low in empathy, a key component of therapeutic alliance. To validate these findings, we will compare content analysis scores with three patient self-reports: perceived therapeutic alliance, perceived empathy in the AI conversation, and baseline empathy typically experienced with their clinicians. Together, these measures will offer a robust evaluation of the therapeutic alliance established by the AI system.
Adherence to recommendations | From enrollment up to 4 months after participation
  Adherence to the recommendations provided by either the structured questionnaire or the conversational AI will be evaluated approximately one month after patient participation. Follow-up includes a structured questionnaire and brief interview, where patients report (1) if they discussed system-generated recommendations with their clinician, and (2) their current medications by direct reference to medication containers. Collected data will allow classification of clinician prescriptions as either concordant or discordant with system-generated recommendations, facilitating evaluation of adherence behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- George Mason University, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data from this study will be shared with the Patient-Centered Outcomes Research Institute (PCORI) and made available through PCORI's designated data repository. Qualified researchers may request access to the data by following PCORI's established data access procedures, which include submission of a research proposal and a signed data use agreement.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available by June 2029, following completion of the final research report, and will remain available for at least 7 years.
Access Criteria: Qualified researchers may request access to de-identified individual participant data and supporting documents (including the protocol, statistical analysis plan, informed consent form, and analytic code) via the PCORI-designated repository. Access to certain data elements may require submission of a research proposal and a signed data use agreement.